CLINICAL TRIAL: NCT06499662
Title: The Influence of Vagus Nerve Neurodynamics on Heart Rate Variability Measured With Sensors in Patients Suffering From Chronic Stress: A Controlled Clinical Trial
Brief Title: Randomised Clinical Trial to Determine the Effect of Vagus Nerve Neurodynamics on the Neurovegetative Nerve System in People With Chronic Stress.
Acronym: VNN-HRV-CCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta de la Plaza (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor-Investigator, Marta de la Plaza, Doctor, European University of Madrid
Organization: European University of Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNNHRV2024-01
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Stress, Psychological Cumulative; Chronic Disease; Heart Rate Variability; Vagal Nerve Stimulation; Autonomic Nervous System Diseases
MeSH Terms: conditions — Stress, Psychological; Chronic Disease; Autonomic Nervous System Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: This study is a controlled clinical trial with a parallel design. Participants will be randomised into two groups: one group will receive a combination of vagus nerve neurodynamics, 6 bpm guided breathing and manual therapy, while the other group will receive only 6 bpm guided breathing and manual therapy. Each group will be treated simultaneously and the results will be compared between groups to assess the effect of neurodynamics on heart rate variability in chronically stressed patients.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study will employ simple blinding. Participants will be blinded to the intervention group to which they belong. Outcome assessors will also be blinded to group assignment to ensure that heart rate variability (HRV) measurements are not influenced by participants' knowledge of the intervention received. Staff delivering interventions will not be blinded due to the nature of neurodynamic and guided breathing techniques, which require knowledge of the specific protocol applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Neurodynamics and Guided Breathing with Manual Therapy (Active Comparator): Participants in this arm will receive a combination of vagus nerve neurodynamics and guided breathing at a rate of 6 breaths per minute (bpm), along with manual therapy. The neurodynamics intervention involves passive movements in the cervical region to enhance vagus nerve function, synchronized with the guided breathing. The manual therapy will include suboccipital inhibition techniques to complement the intervention. The total duration of the intervention will be 15 minutes.
  Interventions: Other: Vagus Nerve Neurodynamics; Other: Guided Breathing; Other: Manual Therapy
- Guided Breathing with Manual Therapy (Active Comparator): Participants in this arm will receive only guided breathing at a rate of 6 breaths per minute (bpm) along with manual therapy. The guided breathing will be diaphragmatic, following a recording that marks the times for inhalation and exhalation. The manual therapy will include suboccipital inhibition techniques applied during the breathing. The total duration of the intervention will be 15 minutes.
  Interventions: Other: Guided Breathing; Other: Manual Therapy

INTERVENTIONS:
Other: Vagus Nerve Neurodynamics — This intervention involves passive cervical movements designed to enhance vagus nerve functionality.
  Arms: Vagus Nerve Neurodynamics and Guided Breathing with Manual Therapy
Other: Guided Breathing — This intervention consists of diaphragmatic breathing guided by a recording to maintain a rate of 6 breaths per minute.
Other: Manual Therapy — This intervention includes suboccipital inhibition techniques applied during the session.

SUMMARY:
This unicentric, controlled clinical trial aims to evaluate the effects of vagus nerve neurodynamics and 6 bpm guided breathing, combined with manual therapy, on heart rate variability (HRV) in patients suffering from chronic stress. A total of 62 participants will be randomly assigned into two groups: one receiving guided breathing and neurodynamics with manual therapy, and the other receiving only guided breathing with manual therapy. HRV will be monitored using Polar® H10 sensors. The primary outcome is the change in HRV, measured pre- and post-intervention. The study is ethically approved by the Hospital Clínico San Carlos.

DETAILED DESCRIPTION:
This unicentric, controlled clinical trial investigates the impact of vagus nerve neurodynamics and guided breathing at a rate of 6 breaths per minute (bpm), in conjunction with manual therapy, on heart rate variability (HRV) in patients with chronic stress.

The study involves 62 participants who will be randomly allocated into two groups. Group 1 will receive a protocol of guided breathing combined with neurodynamics and manual therapy, while Group 2 will follow a protocol of guided breathing with manual therapy only.

Each participant will undergo a 15-minute intervention session where HRV will be continuously monitored using Polar® H10 sensors. The intervention will include guided diaphragmatic breathing at 6 bpm to standardize the respiratory rate across participants, ensuring that HRV measurements reflect the effects of neurodynamics rather than respiratory variations.

The neurodynamics technique involves passive movements in the cervical region to enhance the functionality of the vagus nerve, potentially influencing HRV. This technique will be applied during the intervention period, with specific movements synchronized with the participants' respiratory cycle.

Prior to the intervention, baseline HRV will be recorded during a 7-minute rest period. Post-intervention HRV measurements will also be taken for 7 minutes while participants remain in a supine position. Data analysis will focus on comparing the HRV changes between the two groups, providing insights into the effectiveness of combining neurodynamics with guided breathing and manual therapy.

The study adheres to ethical guidelines and has received approval from the Medical Research Ethics Committee of Hospital Clínico San Carlos

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older.
* Self-perceived chronic stress for at least six months.
* Willingness to provide informed consent and comply with the study procedures

Exclusion Criteria:

* Consumption of tea, caffeine, energy drinks, alcohol, or tobacco within two hours prior to the study.
* Significant neck pain or headache.
* Carotid sinus syndrome.
* Pregnancy.
* Recent cervical or cardiac surgery.
* Recent significant trauma.
* Cancer.
* Neurological disorders affecting muscle tone.
* Underlying conditions such as diabetes mellitus or arterial hypertension.
* Use of beta-blockers.
* Arrhythmias or other cardiac diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) | From the start of the study until 7 minutes post-intervention.
  The primary outcome measure is the change in heart rate variability (HRV) from baseline to post-intervention. HRV will be measured using a Polar® H10 sensor band placed on the participants' chest. HRV data will be recorded during a 7-minute period before the intervention (at rest), during the 15-minute intervention, and during a 7-minute period after the intervention (at rest). Specific HRV parameters to be analyzed include RMSSD (Root Mean Square of the Successive Differences), pNN50 (percentage of adjacent NN intervals that differ by more than 50 ms), and high-frequency power (HF power).

CONTACTS AND LOCATIONS:
Locations (1):
- Marta de la plaza, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No